CLINICAL TRIAL: NCT06293352
Title: Durable, Real-component Antibiotic Spacers Vs All-cement Articulating Spacers for the Treatment of Periprosthetic Knee Infection
Brief Title: Real-component Vs All-cement Articulating Spacers for Periprosthetic Knee Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Adam Edelstein, Assistant Professor of Orthopaedic Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00220012
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Prosthetic-joint Infection; Knee Infection; Arthroplasty Complications; Joint Infection; Arthroplasty, Replacement, Knee
Keywords: randomized trial; patient-reported outcomes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- All-cement articulating spacer (Active Comparator): An articulating spacer with a tibial and femoral component made of cement using molds, that are cemented in place; use of highdose antibiotic cement (at least 2g/batch, including vancomycin and tobramycin); use of dowels at discretion of surgeon; 6 weeks IV antibiotics; intent to reimplant definitive prosthesis if infection eradicated.
  Interventions: Device: All-cement articulating spacer
- Durable, real-component articulating spacer (Active Comparator): Uses metal (or ceramicized metal) on plastic for bearing surface; use of high-dose antibiotic cement (at least 2g/batch, including vancomycin and tobramycin); no cones/sleeves, no pressurized cement in canal; use of stems/dowels/augments and level of constraint at discretion of surgeon; 6 weeks IV antibiotics; intent to leave in situ indefinitely/until clinical failure.
  Interventions: Device: Durable, real-component articulating spacer
- Observation (Other): Patients who do not wish to be randomized or who meet the randomization-specific exclusion criteria will be offered enrolment into the non-randomized, prospective observational arm of the study. The participant and their surgeon will collaboratively decide which of the 2 treatments the participant will receive.
  Interventions: Device: All-cement articulating spacer; Device: Durable, real-component articulating spacer; Device: Rigid Spacer

INTERVENTIONS:
Device: All-cement articulating spacer — Two-stage intervention
  Arms: All-cement articulating spacer; Observation
Device: Durable, real-component articulating spacer — Single stage intervention
  Arms: Durable, real-component articulating spacer; Observation
Device: Rigid Spacer — Observation intervention
  Arms: Observation

SUMMARY:
In the US, if an infection in an artificial knee joint doesn't heal with antibiotics alone, the standard treatment is a two-stage revision of the artificial knee. In the first stage, the surgeon will remove the artificial knee and clean out the area around the knee. They will then place an antibiotic spacer. An antibiotic spacer is a type of artificial joint that will release antibiotics into the knee space continuously over time. The spacer allows only very basic function of the knee. The patient may need to use crutches or a walker while the antibiotic spacer is in place. After surgery to place the antibiotic spacer, the surgeon may prescribe a course of antibiotics as well. Because the antibiotic spacer is not as durable as a regular artificial joint, after the infection is gone, another surgery is required to take the spacer out and put a new artificial knee joint in.

There is another way for artificial joint infections to be treated. This is a one-stage revision. In this treatment, the surgeon will remove the artificial knee and clean out the area around the knee. Then the surgeon will place a new artificial knee in using a special kind of cement that contains antibiotics. The cement will release antibiotics into the knee space continuously over time (the surgeon may prescribe a course of antibiotics as well). The new artificial joint with antibiotic cement will function almost the same as the original artificial knee. This means that while the infection is healing the patient will be able to do most of the regular daily activities. However, the antibiotic cement is not as durable as what is normally used to implant an artificial knee. The artificial knee with the antibiotic cement may need to be replaced with a regular artificial knee. When replacement will need to be done is dependent on patient weight, bone strength and activity level, among other things. When it is time to replace the antibiotic cement artificial knee, the patient will have another surgery where the surgeon will take the antibiotic cement artificial knee and put a new artificial knee joint in.

Investigators know that both the one- and two-stage revision work equally well to heal the infection, but investigators don't know which patients prefer or which provides better function after many years. This study will randomly assign patients to receive either a one-stage or two-stage revision and then follow them for 5 years to ask them about pain, function, and satisfaction.

DETAILED DESCRIPTION:
This study compares to currently used treatments for chronic peri-prosthetic joint infections: Treatment with an all-cement articulating spacer and treatment with a durable, real-component articulating spacer.

An all-cement articulating spacer will be defined as follows: An articulating spacer with a tibial and femoral component made of cement using molds, that are cemented in place; use of high-dose antibiotic cement (at least 2g/batch, including vancomycin and tobramycin); use of dowels at discretion of surgeon; 6 weeks IV antibiotics; intent to reimplant definitive prosthesis if infection eradicated.

A durable, real-component articulating spacer will be defined as follows: Uses metal (or ceramicized metal) on plastic for bearing surface; use of high-dose antibiotic cement (at least 2g/batch, including vancomycin and tobramycin); no cones/sleeves, no pressurized cement in canal; use of stems/dowels/augments and level of constraint at discretion of surgeon; 6 weeks IV antibiotics; intent to leave in situ indefinitely/until clinical failure.

This will be a study with 2 cohorts. We will have a randomized cohort, as well as a nonrandomized prospective observational cohort.

Surgery will be performed by current treatment guidelines in the same manner as if the patient was not in a research study.

All questionnaires will be administered via iPad/online.

The questionnaires administered at the preoperative appointment will consist preoperative patient-reported outcomes (PROs). The preoperative PROs will be determined utilizing PROMIS questionnaires including PROMI-10 Survey and the Knee Injury and Osteoarthritis Outcome - Joint Replacement Score (KOOS-JR), In addition, patient demographic characteristics will be collected including age, sex, race, education and insurance status as well as self-reported comorbidity data.

The questionnaires will be administered again at the 6-week and 6-month, 12-month, and 24- month postoperative time points. In addition, the PROMIS depression scale will be collected at 6 weeks.

The presence and absence any complications, along with complication severity as determined by the PI, during the procedure or during recovery will be extracted from the EMR by the PI and/or Co-investigator after surgery and after every postoperative visit through the 24-month visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a chronic periprosthetic joint infection after a primary total knee arthroplasty with plan for explant and placement of an antibiotic spacer
* PJI defined according to Musculoskeletal Infection Society (MSIS) 2018 Consensus Criteria

Exclusion Criteria:

* Patients who are unable to consent
* Infection at site of revision TKA
* Soft tissue envelope compromise
* Allergies to study materials (cement, vancomycin, tobramycin)
* Incompetent extensor mechanism
* Extensive bone loss

Randomization-specific exclusion criteria

* Extensive soft tissue defect
* Extensor mechanism compromise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
24 month Knee Injury and Osteoarthritis Outcome - Joint Replacement Score (KOOS-JR) | 24 months after surgery
  Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.

SECONDARY OUTCOMES:
24 month 10-item PROMIS Global Health survey (PROMIS-10) | 24 months after surgery
  Raw PROMIS-10 (v1.0) scores for Physical Health (PH) and Mental Health (MH) will be converted to standardized T-score values. A T-score of 50 represents the mean of the general population and higher scores indicate better physical or mental health.

OTHER OUTCOMES:
Revision/reoperation for infection incidence (defined by positive culture by MSIS criteria) | 24 months after surgery
  Count of occurrence of revision/reoperation for infection
Revision/reoperation for infection proportion (defined by positive culture by MSIS criteria) | 24 months after surgery
  Percentage of occurrence of revision/reoperation for infection
Revision for aseptic failure incidence (defined by negative culture by MSIS criteria) | 24 months after surgery
  Count of occurrence of reoperation for aseptic failure
Revision for aseptic failure proportion (defined by negative culture by MSIS criteria) | 24 months after surgery
  Percentage of occurrence of reoperation for aseptic failure

CONTACTS AND LOCATIONS:
Overall Officials: Adam I Edelstein, MD, Principal Investigator — Assistant Professor of Orthopaedic Surgery
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Open to data sharing by request.
Supporting Information: Study Protocol, SAP
Time Frame: Data available after publication of final publication.
Access Criteria: By request.

REFERENCES:
- [Background] Parvizi J, Tan TL, Goswami K, Higuera C, Della Valle C, Chen AF, Shohat N. The 2018 Definition of Periprosthetic Hip and Knee Infection: An Evidence-Based and Validated Criteria. J Arthroplasty. 2018 May;33(5):1309-1314.e2. doi: 10.1016/j.arth.2018.02.078. Epub 2018 Feb 26. PMID 29551303